CLINICAL TRIAL: NCT04035811
Title: Prospective Clinical Assessment Study in Children With Achondroplasia: The PROPEL Trial
Brief Title: Prospective Clinical Assessment Study in Children With Achondroplasia (ACH)
Status: Active, not recruiting | Type: Observational
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Other Study IDs: QBGJ398-001
Record Dates: First submitted 2019-07-20; First posted 2019-07-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Achondroplasia
Keywords: Skeletal dysplasia; Endochondral ossification; Achondroplasia (ACH); Shortened proximal limbs; Fibroblast growth factor receptor 3; FGFR3; Endochondral bone formation; Short-limb disproportionate dwarfism; Quality of life in achondroplasia; Dwarfism; Bone diseases; Musculoskeletal diseases; Osteochondrodysplasia; Genetic diseases; Inborn; Functional abilities; Average growth velocity; Average height velocity; growth; Congenital
MeSH Terms: conditions — Achondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect blood for central assessment of blood biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a long-term, multi-center, observational study in children 2.5 to <17 years with achondroplasia (ACH). The objective is to evaluate growth, ACH-related medical complications, assessments of health-related quality of life, body pain, functional abilities, cognitive functions, and treatments of study participants. No study medication will be administered.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent by study participant or parent(s) or legally authorized representative (LAR) and signed informed assent by the study participant (when applicable)
* Aged 2.5 to <17 years at study entry
* Diagnosis of ACH
* Study participants and parent(s) or LAR(s) are willing and able to comply with study visits and study procedures

Key Exclusion Criteria:

* Have hypochondroplasia or short stature condition other than ACH (e.g. trisomy 21, pseudoachondroplasia, psychosocial short stature)
* In females, having had their menarche
* Height < -2 or > +2 standard deviations for age and sex based on reference tables on growth in children with ACH
* Annualized height growth velocity ≤1.5 cm/year over a period ≥6 months prior to screening
* Current evidence of corneal or retinal disorder/keratopathy
* Current evidence of endocrine alterations of calcium/phosphorus homeostasis
* Have a concurrent disease or condition that in the view of the Investigator and/or Sponsor, may impact growth or where the treatment is known to impact growth.
* Significant abnormality in screening laboratory results.
* Have been treated with growth hormone, insulin-like growth factor 1 (IGF 1), or anabolic steroids in the previous 6 months or long-term treatment (>3 months) at any time
* Have had regular long-term treatment (>1 month) with oral corticosteroids (low-dose ongoing inhaled steroid for asthma is acceptable)
* Have had previous guided growth surgery or limb-lengthening surgery within 12 months prior to screening.

Ages: 30 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with achondroplasia
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Annualized height velocity (cm/year) | Up to 2 years

OTHER OUTCOMES:
Change from baseline in height Z score | Up to 2 years
Change from baseline in upper to lower body ratio (cm) | Up to 2 years
Change from baseline in upper arm to forearm ratio (cm) | Up to 2 years
Change from baseline in upper leg to lower leg ratio (cm) | Up to 2 years
Bone biomarkers (blood) | Up to 2 years
ACH-related NT-AEs | Up to 2 years
ACH-related surgical procedures | Up to 2 years
Changes in health-related quality of life as assessed by Pediatric Quality of Life Inventory (PedsQoL) | Up to 2 years
Changes in health-related quality of life as assessed by Quality of Life in Short Stature Youth questionnaire (QoLISSY) | Up to 2 years
Changes in overall body pain as assessed by Numeric Rating Scale for pain (Pain-NRS) | Up to 2 years
Changes in functional abilities as evaluated by Functional Independence Measure for Children (WeeFIM) | Up to 2 years
Change in psychomotor function assessed by age-appropriate computerized tests (Detection Test) | Up to 2 years
Change in attention assessed by age-appropriate computerized tests (Identification Test) | Up to 2 years
Change in visual learning assessed by age-appropriate computerized tests (One Card Learning Test) | Up to 2 years
Change in working memory assessed by age-appropriate computerized tests (One Back Test) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: QED Therapeutics, Inc. VP, Clinical Development, Study Director — QED Therapeutics
Locations (32):
- United States (8):
  - Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Madison - Waisman Center Bone Dysplasia Clinic, Madison, Wisconsin
- Hospital de Pediatría SAMIC Prof. Dr. Juan P. Garrahan, Buenos Aires, Argentina
- Murdoch Children's Research Institute, Parkville, Australia
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital - London Health Sciences Center, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - University of Montreal, Montreal, Quebec
- France (3):
  - Hopital Femme Mere Enfant, Lyon
  - Hopital Necker-Enfants Malades, Paris
  - Hopital des Enfants, Toulouse
- Otto-von-Guericke-University Magdeburg Medical Fakulty, Magdeburg, Germany
- Italy (2):
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlino, Milan
  - Rare Disease Unit Fondazione Policlinico A Gemelli IRCCS, Rome
- Norway (2):
  - Haukeland Universitetssjukehus, Bergen
  - Oslo Universitetssykehus, Oslo
- KK Women's and Children's Hospital, Singapore, Singapore
- Spain (3):
  - Vithas Hospital San Jose, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- United Kingdom (6):
  - Bristol Royal Hospital for Children, Bristol, England
  - Birmingham Children's Hospital, Birmingham
  - Queen Elizabeth University Hospital, Glasgow
  - St. Thomas' Hospital, London
  - Manchester University Children's Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savarirayan R, De Bergua JM, Arundel P, McDevitt H, Cormier-Daire V, Saraff V, Skae M, Delgado B, Leiva-Gea A, Santos-Simarro F, Salles JP, Nicolino M, Rossi M, Kannu P, Bober MB, Phillips J 3rd, Saal H, Harmatz P, Burren C, Gotway G, Cho T, Muslimova E, Weng R, Rogoff D, Hoover-Fong J, Irving M. Infigratinib in children with achondroplasia: the PROPEL and PROPEL 2 studies. Ther Adv Musculoskelet Dis. 2022 Mar 21;14:1759720X221084848. doi: 10.1177/1759720X221084848. eCollection 2022. PMID 35342457
- See also: Related Info — http://www.QEDtx.com